CLINICAL TRIAL: NCT05086003
Title: Combined Kidney and Hematopoietic Stem Cell Transplantation for Tolerance Induction Between Matched Sibling Donor-recipient Pairs
Brief Title: Combined Kidney and Hematopoietic Stem Cell Transplantation for Tolerance Induction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, moshe yeshurun, Dr Moshe Yeshurun, Head Bone Marrow Unit, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0759-15
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Renal Transplantation
Keywords: Renal transplantation; Bone marrow transplantation; Immune tolerance; Immunosuppression
MeSH Terms: interventions — Bone Marrow Transplantation

STUDY DESIGN:
Intervention Model Description: Combined kidney and bone marrow transplantation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kidney and bone marrow transplantation (Experimental): Combined kidney and bone marrow transplantation after preparation with thymoglobuline and total lymphoid irradiation
  Interventions: Combination Product: Combined kidney and bone marrow transplantation

INTERVENTIONS:
Combination Product: Combined kidney and bone marrow transplantation — Combined kidney and bone marrow transplantation

SUMMARY:
Combined transplantation of kidney and bone marrow between HLA-matched sibling donor-recipient pairs to induce immune tolerance in order to enable complete discontinuation of immunosuppressive therapy without kidney rejection. Hematopoietic stem cells are collected from the donor 4 to 8 weeks before kidney transplantation, CD34 cells are enriched by positive selection and cryopreserved. The day after kidney transplantation the recipient starts conditioning therapy with thymoglobuline, total lymphoid irradiation, steroids, tacrolimus and mycophenolate mofetil. Eleven days after kidney transplantation the stem cell graft is thawed and infused to the recipient. If mixed donor chimerism is successfully maintained more than 6 months without rejection, then immunosuppression may be tapered off until complete discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* Matched siblings
* No contra-indication to thymoglobuline or total lymphoid irradiation

Exclusion Criteria:

* Pregnant women or breast feeding
* Infection with HIV, HBV or HCV
* Previous or presnt malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-01-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of transplanted patients who were able to discontinue immunosuppression 12 months after transplantation. | 12 months
  Proportion of transplanted patients who were able to discontinue immunosuppression 12 months after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Yeshurun, MD, Principal Investigator — Institution of Hematology, Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No